CLINICAL TRIAL: NCT03845283
Title: Optimization and Evaluation of a Tailored Behavioral eHealth/mHealth Weight Loss Intervention for Cardiac Rehabilitation Patients Using the Multiphase Optimization Strategy
Brief Title: Creating an Optimized Technology-Based Weight Loss Program for Cardiac Rehabilitation Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: K23HL136845 (NIH); K23HL136845 (NIH)
Record Dates: First submitted 2019-02-05; First posted 2019-02-19 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases; Obesity
Keywords: Cardiovascular Diseases; Obesity; Multiphase Optimization Strategy; Technology; Weight Loss; Cardiac Rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Physical Activity (Experimental): Participants will receive the core 6-month weight loss program and the tailored intervention to promote structured physical activity.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Physical Activity Intervention
- Core Program (Experimental): Participants will receive the core 6-month weight loss program alone. This program includes weekly lessons for the first 12 weeks and monthly lessons for the remaining 12 weeks. Participants will track their intake, physical activity, and weight, input these data into the system, and received tailored feedback.
  Interventions: Behavioral: Online Behavioral Weight Loss Program
- Physical Activity & Virtual Meetings (Experimental): Participants will receive the core 6-month weight loss program, the tailored intervention to promote structured physical activity, and the virtual meetings to support weight loss.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Physical Activity Intervention; Behavioral: Virtual Meetings
- Virtual Meetings (Experimental): Participants will receive the core 6-month weight loss program and the virtual meetings to support weight loss.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Meetings
- Physical Activity & Virtual Reality (Experimental): Participants will receive the core 6-month weight loss program, the tailored intervention to promote structured physical activity, and access to the virtual reality platform for behavioral weight loss skills training.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Physical Activity Intervention; Behavioral: Virtual Reality
- Virtual Reality (Experimental): Participants will receive the core 6-month weight loss program and access to the virtual reality platform for behavioral weight loss skills training.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality
- Physical Activity, Virtual Reality, & Virtual Meetings (Experimental): Participants will receive the core 6-month weight loss program, the tailored intervention to promote structured physical activity, the virtual meetings to support weight loss, and access to the virtual reality platform for behavioral weight loss skills training.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Physical Activity Intervention; Behavioral: Virtual Reality; Behavioral: Virtual Meetings
- Virtual Reality & Virtual Meetings (Experimental): Participants will receive the core 6-month weight loss program, access to the virtual reality platform for behavioral weight loss skills training, and the virtual meetings to support weight loss.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality; Behavioral: Virtual Meetings
- Physical Activity & Bite Counter (Experimental): Participants will receive the core 6-month weight loss program, the tailored intervention to promote structured physical activity, and the Bite Counter device to reduce dietary intake.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Physical Activity Intervention; Behavioral: Bite Counter
- Bite Counter (Experimental): Participants will receive the core 6-month weight loss program and the Bite Counter device to reduce dietary intake.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Bite Counter
- Physical Activity, Bite Counter, & Virtual Meetings (Experimental): Participants will receive the core 6-month weight loss program, the tailored intervention to promote structured physical activity, the Bite Counter device to reduce dietary intake, and the virtual meetings to support weight loss.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Physical Activity Intervention; Behavioral: Bite Counter; Behavioral: Virtual Meetings
- Bite Counter & Virtual Meetings (Experimental): Participants will receive the core 6-month weight loss program, the Bite Counter device to reduce dietary intake, and the virtual meetings to support weight loss.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Bite Counter; Behavioral: Virtual Meetings
- Physical Activity, Bite Counter, & Virtual Reality (Experimental): Participants will receive the core 6-month weight loss program, the tailored intervention to promote structured physical activity, the Bite Counter device to reduce dietary intake, and access to the virtual reality platform for behavioral weight loss skills training.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Physical Activity Intervention; Behavioral: Bite Counter; Behavioral: Virtual Reality
- Bite Counter & Virtual Reality (Experimental): Participants will receive the core 6-month weight loss program, the Bite Counter device to reduce dietary intake, and access to the virtual reality platform for behavioral weight loss skills training.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Bite Counter; Behavioral: Virtual Reality
- Physical Activity, Bite Counter, Virtual Reality & Meetings (Experimental): Participants will receive the core 6-month weight loss program, the tailored intervention to promote structured physical activity, the Bite Counter device to reduce dietary intake, access to the virtual reality platform for behavioral weight loss skills training, and the virtual meetings to support weight loss.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Physical Activity Intervention; Behavioral: Bite Counter; Behavioral: Virtual Reality; Behavioral: Virtual Meetings
- Bite Counter, Virtual Reality, & Virtual Meetings (Experimental): Participants will receive the core 6-month weight loss program, the Bite Counter device to reduce dietary intake, access to the virtual reality platform for behavioral weight loss skills training, and the virtual meetings to support weight loss.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Bite Counter; Behavioral: Virtual Reality; Behavioral: Virtual Meetings

INTERVENTIONS:
Behavioral: Online Behavioral Weight Loss Program — A self-guided, online program that helps participants reduce excess calories and gradually increase physical activity.
Behavioral: Physical Activity Intervention — An program designed to help participants gradually increase their physical activity and maintain an active lifestyle. The program encourages bouts of moderate-to-vigorous physical activity. Participants in this group will receive a Fitbit Versa to help them monitor their physical activity that they will be advised to wear daily. Participants will receive brief (5-10 minute) lessons weekly for the first 3 months and monthly for the last 3 months.
  Arms: Physical Activity; Physical Activity & Bite Counter; Physical Activity & Virtual Meetings; Physical Activity & Virtual Reality; Physical Activity, Bite Counter, & Virtual Meetings; Physical Activity, Bite Counter, & Virtual Reality; Physical Activity, Bite Counter, Virtual Reality & Meetings; Physical Activity, Virtual Reality, & Virtual Meetings
Behavioral: Bite Counter — Participants will receive a Bite Counter device to help them monitor and reduce their within-meal consumption. Participants will be asked to wear the device daily.
  Arms: Bite Counter; Bite Counter & Virtual Meetings; Bite Counter & Virtual Reality; Bite Counter, Virtual Reality, & Virtual Meetings; Physical Activity & Bite Counter; Physical Activity, Bite Counter, & Virtual Meetings; Physical Activity, Bite Counter, & Virtual Reality; Physical Activity, Bite Counter, Virtual Reality & Meetings
Behavioral: Virtual Reality — This program allows participants to practice behavioral weight loss skills using a virtual reality system compatible with their home device. This program helps patients practice these skills in the following artificial settings: at home, at work, at the gym, and at a party. Each participant will be asked to play through each scene at least once during their participation, though they are encouraged to use the program regularly.
  Arms: Bite Counter & Virtual Reality; Bite Counter, Virtual Reality, & Virtual Meetings; Physical Activity & Virtual Reality; Physical Activity, Bite Counter, & Virtual Reality; Physical Activity, Bite Counter, Virtual Reality & Meetings; Physical Activity, Virtual Reality, & Virtual Meetings; Virtual Reality; Virtual Reality & Virtual Meetings
Behavioral: Virtual Meetings — Participants will attend virtual meetings using their own device. Each virtual meeting focuses on a specific topic that will help patients lose weight. Participants are asked to virtually attend at least 6 meetings during their participation. There is no limit to how many they can attend. The meeting topics will rotate and repeat on a schedule.
  Arms: Bite Counter & Virtual Meetings; Bite Counter, Virtual Reality, & Virtual Meetings; Physical Activity & Virtual Meetings; Physical Activity, Bite Counter, & Virtual Meetings; Physical Activity, Bite Counter, Virtual Reality & Meetings; Physical Activity, Virtual Reality, & Virtual Meetings; Virtual Meetings; Virtual Reality & Virtual Meetings

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the United States. Cardiac rehabilitation (CR) is the main treatment for heart attacks and other types of CVD. It is based on science, it saves money, and it is widely-available. Each session (of which there are a few each week for 3 months) combines supervised exercise and instruction. The goals are to improve overall health and reduce cardiovascular risk in individuals with established CVD. CR produces almost no weight loss (WL); if a person has excess weight while in CR (the majority of participants have overweight or obesity), losing weight could really reduce their risk of having another heart attack. The best treatment available for weight loss, in-person behavioral weight loss interventions (BWLs), produce enough WL that they improve health and disease risk/severity. However, in-person BWLs are too much work to be carried out in CR. A previous fully automated 3-month online program, Rx Weight Loss (RxWL), produced good WL in many different settings. Dr. Goldstein aims to tailor RxWL for use in CR. The study will use the Multiphase Optimization Strategy (MOST) to test innovative eHealth/mHealth intervention components that might work well for people when combined with RxWL. The study will include 160 patients (each randomized to receive 0-4 of the components). The components are: (a) a Fitbit with a goal-setting program; (b) a bite counting device; (c) a Web-based virtual reality (VR) intervention ; and (d) virtual meetings. By the 6-month follow-up, the investigators will know if any of those 4 components helped people lose more weight. If a component produced at least 2% WL, it will be studied further by being included in a new intervention to be tested in the next study.

ELIGIBILITY:
Inclusion Criteria:

* currently a participant in The Miriam Hospital's or Newport Hospital's outpatient phase II cardiac rehabilitation program
* medical clearance to participate by the Medical Director
* a body mass index (BMI) between 27-45 kg/m2
* must have a personal computer in their home with internet access
* must read and understand English
* willing to use technology to assist with weight loss

Exclusion Criteria:

* currently in another weight loss program
* taking weight loss medication
* weight loss of ≥ 5% of body weight in the past 6 months
* currently pregnant, lactating, < 6 months post-partum, or plans to become pregnant during the next year
* report of loss of consciousness on the Physical Activity Readiness Questionnaire
* New York Heart Association Class IV heart failure
* heart transplant in the last 3 months
* receipt of left ventricular assist device in the last 2 months
* a physician diagnosis of dementia
* a physician prescription for 24 hours of oxygen therapy daily
* coronary artery bypass surgery in the last 4 weeks
* current participation in dialysis
* inability to walk 1 block without stopping
* report of conditions that in the opinion of the investigators would render them potentially unlikely to follow the protocol including terminal illness, substance abuse, eating disorder, or other significant psychiatric problems

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Weight Change | At baseline, 3-, and 6-months after initiating the program
  The difference between initial weight and weight at the follow-up assessments. Patients will be asked to step on a scale at the assessment clinic.

SECONDARY OUTCOMES:
Structured Weekly Moderate-to-Vigorous Physical Activity Minutes | At baseline, 3-, and 6-months after initiating the program
  Structured MVPA minutes will be measured via a SenseWear Armband monitor (BodyMedia, Inc, Pittsburgh PA, USA). This multi-sensor monitor worn on the upper triceps wirelessly integrates motion data from a triaxial accelerometer with other sensors to estimate energy expenditure and activity intensity. Everyone will be asked to wear the armband during waking hours across the 7-day period prior to each assessment. Participants will be required to provide at least 5 days of data (including 1 weekend day), defined as ≥ 600 min during the hours of 7 am to 11 pm, to be included in analyses.
Number of Bites | At baseline, 3-, and 6-months after initiating the program
  All study participants' average number of recorded daily bites of food over 7 consecutive days will be assessed by a Bite Counter (Bite Technologies, Pendleton SC, USA) with the display inactivated. Participants' average number of daily bites will be compared from each 7-day period prior to each assessment.
Weight Control Practices | At baseline, 3-, and 6-months after initiating the program
  The validated, widely-used Weight Control Practices Scale measures the health behaviors an individual executes to influence energy balance and is targeted by the VR program. All participants will complete this measure at each assessment point. The overall scale scores range from 0-30 where higher scores indicate that the participant is using more strategies to control their weight. The subscale scores, which assess dietary choices (score range 0-10), self-monitoring strategies (score range 0-8), physical activity (score range 0-6), and psychological coping (score range 0-7), will also be examined. Higher scores on the subscales indicate greater weight control (which is a better outcome). Subscale scores are summed to compute the total scale score.
Weight Loss Self-Efficacy: Weight Efficacy Lifestyle Questionnaire | At baseline, 3-, and 6-months after initiating the program
  This is the participant's confidence in implementing BWL skills. It will be targeted by the virtual meetings and will be measured via the well-validated Weight Efficacy Lifestyle Questionnaire in all participants. The scores can range from 0-180 where higher scores indicate more weight loss self-efficacy and better outcomes.

OTHER OUTCOMES:
Overall Behavioral Self-Management in Cardiac Rehabilitation | At baseline, 3-, and 6-months after initiating the program
  All participants will complete a newly-developed self-management inventory designed specifically for cardiac rehabilitation patients. The total score can range from 54-300, with higher scores generally reflecting better self-management.

CONTACTS AND LOCATIONS:
Locations (1):
- The Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided
The raw data from the current project are too large to easily transfer to individual investigators. As such, the investigators plan to develop a cost-effective, safe plan for sharing de-identified participant data upon reasonable request by other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT03845283/ICF_001.pdf